CLINICAL TRIAL: NCT02447367
Title: Randomized, Open-label, Single Dose, Two-way Crossover, Clinical Trial to Investigate the Effect of Food on the Pharmacokinetic of JLP-1207 After Oral Administration in Healthy Male Volunteers
Brief Title: Investigate the Effect of Food on the Pharmacokinetic of JLP-1207 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1207-P1-FE
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-06

CONDITIONS: LUTS; Benign Prostatic Hyperplasia; Overactive Bladder
Keywords: α1-blockers; antimuscarinic agent
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- JLP-1207, Fasted followed by fed (Experimental): JLP-1207 dosing in the fasted state followed by fed dosing
  Interventions: Drug: JLP-1207(Fasted)
- JLP-1207, Fed followed by fasted (Experimental): JLP-1207 dosing in the fed state followed by fasted dosing
  Interventions: Drug: JLP-1207(Fed)

INTERVENTIONS:
Drug: JLP-1207(Fasted) — Fasted followed by fed in period 1, the subjects will receive an oral pill of JLP-1207 under fasted condition.
  Arms: JLP-1207, Fasted followed by fed
Drug: JLP-1207(Fed) — Fed followed by fasted in period 1, the subjects will receive an oral pill of JLP-1207 under fed condition
  Arms: JLP-1207, Fed followed by fasted

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic drug interaction between Solifenacin and Tamsulosin in healthy male volunteers.

DETAILED DESCRIPTION:
A randomized, open-label, single dose, two-way crossover study

ELIGIBILITY:
Inclusion Criteria:

* 19~45 years healthy male
* Body weight is over 55kg, BMI measurement 18.0kg/m^2~ 27.0kg/m^2
* Signed informed consent form from to participate voluntarily and to comply with the trial requirements.
* Researchers determined suitable volunteers through physical examination, laboratory tests

Exclusion Criteria:

* History of clinically significant liver, kidneys, nervous system, immune system, respiratory, endocrine disorders or tumor or blood disorders, cardiovascular diseases, mental disorders (mood disorders, obsessive-compulsive disorder, etc.)
* Sitting SBP>150mmHg or <100mmHg, sitting DBP>100mmHg or <60mmHg, after 3 minutes break
* An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
* Have a gastrointestinal disease history that can affect drug absorption (Crohn's disease ulcers, etc) or surgery (except simple appendectomy or hernia surgery)
* History of drug abuse
* Positive urine drug screening
* Administrated investigational product in a previous clinical trial within 90 days of the first administration day in this study.
* Donated blood within 60 days prior to the first administration day in this study.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUClast, Cmax, AUCinf | 192 hours

SECONDARY OUTCOMES:
Tmax | 192 hours
t1/2 | 192 hours
CL/F | 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital(SNUH)

IPD SHARING:
Plan to Share IPD: No